CLINICAL TRIAL: NCT06085625
Title: A Randomized Control Trial for Patient Reported Outcomes and Safety in Outpatient Thyroid Lobectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0511; NCI-2023-08793 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Thyroid Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Reported Outcomes and Safety in Outpatient Thyroid Lobectomy (Experimental): Participants will first complete a survey about the severity of your symptoms. This will be done at your pre-surgery (pre-operative) visit and should take about 5-10 minutes to complete.
  Study Groups
  At your pre-surgery visit, you will be assigned to either be sent home on the same day as surgery or to stay in the hospital overnight (or longer) for observation. This will be determined based on which group your surgeon has been assigned to. Participants will be told which group you are in.
  Interventions: Behavioral: Pre-Surgery Survey; Behavioral: Post-Surgery Surveys

INTERVENTIONS:
Behavioral: Pre-Surgery Survey — Participants will be asked to complete a survey 3 times (before surgery, after surgery, and 2 weeks after surgery). You will be monitored for up to 1 month after your surgery, where you may be contacted by a study provider virtually or in person to ask you about medication usage and heath care needs.
Behavioral: Post-Surgery Surveys — After surgery, Participants will complete the same survey as in the pre-surgery visit about 1 day and then 2 weeks after surgery. These surveys will be completed electronically through the MyChart system. They will take about 5-10 minutes to complete and must be done within 24 hours after receiving the survey.
  Participants will be monitored for 1 month after your surgery, including your standard-of-care postoperative visit at about 2 weeks. You may be contacted by a provider for a phone or in person visit at the 1-month time point to ask how you are doing.

SUMMARY:
To compare same-day discharge and overnight (or longer) observation practices and learn more about the differences in patient preferences, safety outcomes, and economic and resource impact

DETAILED DESCRIPTION:
Primary Objective:

--To determine whether same-day discharge is non-inferior to usual care (overnight stay) with regard to the MD Anderson Symptom Inventory - Thyroid (MDASI-Thyroid) mean severity score, as assessed at 2 weeks post-procedure in patients undergoing thyroid lobectomy.

Secondary Objectives:

* To determine whether same-day discharge is non-inferior to usual care (overnight stay) with regard to the MDASI-Thyroid mean severity score, as assessed at 24 hours post-procedure in patients undergoing thyroid lobectomy.
* To determine whether the two arms differ by incidence of deviations from normal as defined by post-operative hematoma, emergency care presentation, readmission/re-intervention, high pain severity scores, and 30-day mortality.
* To determine whether morphine milligram equivalents (MME) used over the 2-week post-operative period differs between patients who receive same-day discharge vs. those who receive usual care (overnight stay) after receiving thyroid lobectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age
2. Patients undergoing initial partial or complete thyroid lobectomy
3. English and non-English speaking patients are eligible

Exclusion Criteria:

1. Increased risk of bleeding (e.g., Aspirin, antiplatelet therapy, or anticoagulation that cannot be held 5 days before surgery, baseline thrombocytopenia <50,000/µL)
2. Pre-existing medical comorbidities or poor performance status (Eastern Cooperative Oncology Group performance status >2) that would otherwise dictate overnight in-hospital postoperative observation
3. Increased distance of residence from index hospital (>50 miles) or inability to stay within the targeted area (<50 miles) postoperatively prohibiting timely return to the index hospital in emergent situations
4. Lives alone or unable to independently perform Activities of Daily Living and no available caregiver in the immediate postoperative period (POD 0-3)
5. Pregnant women will not be included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Graham, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org